CLINICAL TRIAL: NCT05926375
Title: Effect of HINEX Jelly on Nutritional Status in People With Possible Sarcopenia or Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University (Other)
Collaborators: Taiwan Otsuka Pharm. Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: N202112052
Record Dates: First submitted 2023-06-19; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-01

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: The experiment lasted for 20 weeks, including 8 weeks self-controlled phase, 8 weeks supplement phase and 4 weeks washout period. In self-controlled phase would intake 400~500 kcal breakfast and in supplement phase consume one servings of jelly high protein supplement with 100~200 kcal food at breakfast. Subjects were randomly divided into "first intervention group" and "post intervention group". The first intervention group used HINEX Jelly as daily breakfast during the first to 8th weeks of the experiment, the 9th to 12th week is the wash out period, the 13th to the 20th week is the selfcontrol period; the post-intervention group is in the first to the 8th week of self-control period,the 9th to 12th week is the wash out period, and the 13th to the 20th week is used HINEX Jelly as daily breakfast, as well as maintained their regular diet and medication, but do exercise lifestyle modification during 20-week experimental period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first intervention group (Supp-Con sequence) (Experimental): The first intervention group used HINEX Jelly as daily breakfast during the first to 8th weeks of the experiment, the 9th to 12th week is the wash out period, the 13th to the 20th week is the selfcontrol period.
  Interventions: Dietary Supplement: HINEX Jelly ( jelly high protein supplement)
- post intervention group (Con-Supp sequence) (Experimental): the post-intervention group is in the first to the 8th week of self-control period,the 9th to 12th week is the wash out period, and the 13th to the 20th week is used HINEX Jelly as daily breakfast.
  Interventions: Dietary Supplement: HINEX Jelly ( jelly high protein supplement)

INTERVENTIONS:
Dietary Supplement: HINEX Jelly ( jelly high protein supplement) — In self-controlled phase,which intake 400~500 kcal breakfast, or in supplement phase consume one servings of jelly high protein supplement (303 kcal, 15 g protein and 2400 mg BCAA per serving) and 100~200 kcal food at breakfast per day, for 8 weeks.

SUMMARY:
HINEX Jelly is a jelly high protein supplement. This report is to investigate whether jelly high protein supplement can achieve greater muscle mass, muscle strength, physical performance and nutritional status in sarcopenia or possible sarcopenia subjects. It is 20 weeks randomized, crossover, self-controlled trials. The screening, recruitment and trial period were carried out from Feb, 2022 to Mar, 2023. Patients were randomized to either a self-controlled phase,which intake 400~500 kcal breakfast, or a supplement phase consume one servings of jelly high protein supplement (303 kcal, 15 g protein and 2400 mg BCAA per serving) and 100~200 kcal food at breakfast per day, for 8 weeks. After a 4-week washout they cross over to the alternate treatment. The anthropometric measurements, sarcopenia parameters, nutritional assessment and hematology assessment data were measured at the week 0,8,12,20 and 24-hour dietary record were recorded at week 1,8,13,20.

DETAILED DESCRIPTION:
Parameters of sarcopenia, including the muscle mass assessment, handgrip strength and physical performance assessment.Muscle mass and body composition were measured by bioelectrical impedance analysis (BIA). A hand dynamometer was used to measure handgrip strength. Physical performance was measured by short physical performance battery (SPPB), 6-meter gait speed and 5-time chair stand test. Mini nutritional assessment (MNA) used to measure nutritional status. The hematology assessment including total protein, albumin, pre-albumin, transferrin, c-reactive protein (CRP), vitamin D, calcium, glucose, insulin, homeostasis model assessment-estimated insulin resistance (HOMA-IR), total cholesterol, triacylglycerol, creatinine, creatine-kinase, alkaline phosphatase, glutamic oxaloacetic transaminase (GOT), glutamic pyruvic transaminase (GPT) and complete blood count.

ELIGIBILITY:
Inclusion Criteria:

* 40-85 years old, middle-aged and elderly subjects with possible sarcopenia or sarcopenia. According to AWGS 2019, possible sarcopenia is defined as (1) handgrip strength < 28 kg in men and < 18 kg in women or (2) 5-time chair stand test ≥ 12 seconds; sarcopenia is defined as meet (1) or (2) plus appendicular skeletal muscle mass index (ASMI) < 7.0 kg/m2 in men and < 5.7 kg/m2 in women.

Exclusion Criteria:

* BMI>35 kg/m2, Taking any special diet (i.e. vegan), be allergic to ingredient (i.e. milk or soy bean) and any seriously acute or chronic lung, liver, kidney, gastrointestinal, cancers diseases history.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-06-28 (Estimated)

PRIMARY OUTCOMES:
muscle mass | week 0,8,12,20
  the change of muscle mass and measured via bioelectrical impedance analysis(BIA)
hand grip strength | week 0,8,12,20
  the change of hand grip strength as the marker of muscle strength.Measured via hand grip dynamometry.
5-time chair stand test | week 0,8,12,20
  the change of 5-time chair stand test as the marker of physical performance.

SECONDARY OUTCOMES:
short physical performance battery | week 0,8,12,20
  the change of short physical performance battery as the marker of physical performance.
6-meter gait speed | week 0,8,12,20
  the change of 6-meter gait speed as the marker of physical performance.
Mini nutritional assessment | week 0,8,12,20
  the change of 6-meter gait speed as the marker of nutritional status.

OTHER OUTCOMES:
General clinical chemistry of blood lipid | week 0,8,12,20
  the change of lipid profile (total cholesterol and triglyceride) and measured via automated clinical chemistry analyzer
General clinical chemistry of blood sugar | week 0,8,12,20
  the change of blood sugar (glucose, insulin) and measured via automated clinical chemistry analyzer. Use the glucose, insulin concentration to calculate homeostasis model assessment-estimated insulin resistance (HOMA-IR).
General clinical chemistry of liver function | week 0,8,12,20
  the change of liver function function ( glutamic oxaloacetic transaminase (GOT), glutamic pyruvic transaminase (GPT)) and measured via automated clinical chemistry analyzer
General clinical chemistry of kidney function | week 0,8,12,20
  the change of liver function and kidney function (creatinine) and measured via automated clinical chemistry analyzer
General clinical chemistry of nutritional status | week 0,8,12,20
  the change of nutritional status (total protein in g/dL, albumin in g/dL, pre-albumin in mg/dL, transferrin in mg/dL) and measured via automated clinical chemistry analyzer
General clinical chemistry of vitamin D status | week 0,8,12,20
  the change of vitamin D status and measured via automated clinical chemistry analyzer
C-reactive protein (CRP) | week 0,8,12,20
  the change of inflammatory marker C-reactive protein (CRP) measured via automated clinical chemistry analyzer
Tumor Necrosis Factor-α(TNF-α) | week 0,8,12,20
  the change of inflammatory marker Tumor Necrosis Factor-α(TNF-α) measured via commercial kit

CONTACTS AND LOCATIONS:
Overall Officials: Jane C-J Chao, Ph.D., Study Chair — Taipei Medical University, Taiwan, R.O.C.
Locations (1):
- Taipei Medical University, New Taipei City, Zhonghe Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No